CLINICAL TRIAL: NCT06393803
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of Single and Multiple Doses of KH607 Tablets in Chinese Healthy Volunteers
Brief Title: Phase 1 Study of KH607 Tablets
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KH607-30101
Record Dates: First submitted 2024-01-04; First posted 2024-05-01 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- KH607 Cohort 1 (Experimental): Subject received a single KH607 tablets dose of 2mg KH607 tablets or matching placebo.
  Interventions: Drug: 2mg KH607 tablets
- KH607 Cohort 2 (Experimental): Subject received a single KH607 tablets dose of 5mg KH607 tablets or matching placebo.
  Interventions: Drug: 5mg KH607 tablets
- KH607 Cohort 3 (Experimental): Subject received a single KH607 tablets dose of 10mg KH607 tablets or matching placebo.
  Interventions: Drug: 10mg KH607 tablets
- KH607 Cohort 4 (Experimental): Subject received a single KH607 tablets dose of 20mg KH607 tablets or matching placebo.
  Interventions: Drug: 20mg KH607 tablets
- KH607 Cohort 5 (Experimental): Subject received a single KH607 tablets dose of 30mg KH607 tablets or matching placebo.
  Interventions: Drug: 30mg KH607 tablets
- KH607 Cohort 6 (Experimental): Subject received a single KH607 tablets dose of 40mg KH607 tablets or matching placebo.
  Interventions: Drug: 40mg KH607 tablets
- KH607 Cohort 7 (Experimental): Subject received a single KH607 tablets dose of 50mg KH607 tablets or matching placebo.
  Interventions: Drug: 50mg KH607 tablets
- KH607 Cohort 8 (Experimental): Subject received a single KH607 tablets dose of 60mg KH607 tablets or matching placebo.
  Interventions: Drug: 60mg KH607 tablets
- KH607 Cohort 9 (Experimental): Subject received 10mg KH607 or matching placebo, oncely daily from Day 1 to Day 7.
  Interventions: Drug: 10mg KH607 tablets
- KH607 Cohort 10 (Experimental): Subjects receive 20mg KH607 or matching placebo, once daily from Day 1 to Day 7.
  Interventions: Drug: 20mg KH607 tablets
- KH607 Cohort 11 (Experimental): Subjects receive 30mg KH607 or matching placebo, once daily from Day 1 to Day 7.
  Interventions: Drug: 30mg KH607 tablets

INTERVENTIONS:
Drug: 2mg KH607 tablets — Subject receive KH607 tablets or placebo orally single dose.
  Arms: KH607 Cohort 1
Drug: 5mg KH607 tablets — Subject receive KH607 tablets or placebo orally single dose.
  Arms: KH607 Cohort 2
Drug: 10mg KH607 tablets — Subject receive KH607 tablets or placebo orally single dose or multiple doses.
  Arms: KH607 Cohort 3; KH607 Cohort 9
Drug: 20mg KH607 tablets — Subject receive KH607 tablets or placebo orally single dose or multiple doses.
  Arms: KH607 Cohort 10; KH607 Cohort 4
Drug: 30mg KH607 tablets — Subject receive KH607 tablets or placebo orally single dose or multiple doses.
  Arms: KH607 Cohort 11; KH607 Cohort 5
Drug: 40mg KH607 tablets — Subject receive KH607 tablets or placebo orally single dose.
  Arms: KH607 Cohort 6
Drug: 50mg KH607 tablets — Subject receive KH607 tablets or placebo orally single dose.
  Arms: KH607 Cohort 7
Drug: 60mg KH607 tablets — Subject receive KH607 tablets or placebo orally single dose.
  Arms: KH607 Cohort 8

SUMMARY:
This study was a single-center, randomized, double-blind, placebo-controlled study divided into a Single Ascending Dose (SAD) stage and a Multiple Ascending Dose (MAD) stage. The primary objective was to evaluate the safety and tolerability of KH607 tablets in Chinese healthy volunteers.

DETAILED DESCRIPTION:
This study consists of two parts: Part 1-SAD phase and Part 2- MAD phase. There will be eight cohorts in Part 1 and three cohorts in Part 2 of this study.

The SAD study will enroll approximately 58 HVs across 8 dose cohorts. The dose cohorts will include the following dose levels: 2 mg, 5 mg, 10 mg, 20 mg, 30 mg, 40 mg, 50mg and 60 mg. All participants in Part 1 will be administered with a single oral dose of KH607 or its matching placebo under fasted condition.

Approximately 30 HVs will be enrolled in the multiple ascending dose study. The dose cohorts will include the following dose levels: 10 mg, 20 mg, 30 mg.At each cohort, 10 subjects will be randomized in a ratio of 8:2 to be receive KH607 or placebo once daily for continuous 7 days (QDx7d) in a double-blind manner.

Additionally, this study will explore the effect of food on the PK of a single oral administration of KH607 in one selected SAD cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, male and female volunteers, 18 to 55 years of age, inclusive.
2. Male weight ≥ 50kg, female weight ≥ 45kg, and body mass index ≥ 19 to ≤ 28 kg/m2 at the screening period.

Exclusion Criteria:

1. Vulnerable groups include the Investigator and his or her immediate family members (spouse, parents, children, siblings), non-immediate family members involved in the study, or individuals who may be participating under coercion or undue influence.
2. Subjects whose C-SSRS suggests that they are at risk for suicide at the screening period, or with the risk for suicide based on the Investigator's clinical judgment, or with a history of suicidal or self-harming behavior.
3. Subjects with SSS ≥3 or MOAA/S ≤4 during the screening period.
4. Subjects with a history of surgery for gastrointestinal disorders or current GI disorders that may interfere with drug absorption, or who have undergone major surgery within the 3 months prior to the screening period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-10-21 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
12-lead ECGs | Screening up to Part 1 Days, Part 2 Day14.
  Using a standard 12-lead ECG machine that automatically calculates heart rate and measures PR interval, RR interval, QRS interval, QT interval and QTc interval. ECGs will be reviewed by the Investigator on an ongoing basis as safety assessments.
Physical Examination | Screening up to Part 1 Days, Part 2 Day14.
12-lead ECGs | Screening up to Part 2 Day14.
  Using a standard 12-lead ECG machine that automatically calculate heart rate and measures PR interval, RR interval, QRS interval, QT interval, QTc interval. ECGs will be reviewed by the Investigator on an ongoing basis as safety assessments.
Stanford Sleepiness Scale | Screening up to Part 1 Day3，Part 2 Day14.
  Participants rate their current sleepiness on a scale of 1 to 7, where scale of 1 indicates feeling active, vital, alert, or wide awake. Scale of 7 indicates no longer fighting sleep, sleep onset soon, and having dream-like thoughts.
Modified Observer's Assessment of Alertness/Sedation scale | Screening up to Part 1 Day3，Part 2 Day14.
  The MOAA/S ranges from 0 to 5, with a score of 5 defined as awake or minimally sedated, and a score of 0 defined as general anaesthesia.

SECONDARY OUTCOMES:
Columbia-Suicide Severity Rating Scale | Screening up to Part 1 Day3，Part 2 Day14.
  The C-SSRS scale consists of three subscales: suicidal ideation, intensity of ideation and suicidal behavior.
Observed maximum plasma concentration (Cmax) | Up to 48 hours after dosing in Part 1.
Time to reach maximum plasma concentration (Tmax) | Up to 48 hours after dosing in Part 1.
Elimination Halflife (T1/2) | Up to 48 hours after dosing in Part 1.
Area under the concentration-time curve from time zero to last time of quantifiable concentration（AUC0-t） | Up to 48 hours after dosing in Part 1.
Apparent Distribution Volume (Vd) | Up to 48 hours after dosing in Part 1.
Apparent Total Plasma Clearance (CL) | Up to 48 hours after dosing in Part 1.
Elimination Rate Constant (Kel) | Up to 48 hours after dosing in Part 1.
Mean Residence Time(MRT) | Up to 48 hours after dosing in Part 1.
Steady-state valley concentration（Css,min） | Up to 24 hours after Day7 dosing in Part 2.
Steady-state peak concentration（Css,max） | Up to 24 hours after Day7 dosing in Part 2.
Mean steady-state blood concentration（Css,av） | Up to 24 hours after Day7 dosing in Part 2.
Steady state area under the curve（AUC0-tau） | Up to 24 hours after Day7 dosing in Part 2.
Accumulation Index（Rac） | Up to 24 hours after Day7 dosing in Part 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anding Hospital Affiliated to Capital Medical University, Beijing, China